CLINICAL TRIAL: NCT05537103
Title: Adolescents Seeking COVID Vaccination
Brief Title: Adolescents Seeking COVID Vaccination (Teen COVID Vax)
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10000982; 000982-CC
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Ease Of Access To Covid Vaccine
Keywords: Survey; Teens; Choices; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: 15-17 year olds from US general population

SUMMARY:
Background:

Information is limited on the experience of children aged 15 to 17 who have or have not been vaccinated against COVID-19. Research has assessed attitudes toward COVID-19 vaccination among adults and parents of teenagers. Few surveys have explored attitudes among teens themselves.

Objective:

This anonymous cross-sectional survey of a national sample US teens to find out about their experiences and attitudes on getting vaccinated for COVID-19. This study will be conducted in collaboration with a national firm (Qualtrics) responsible for the recruitment and data collection.

Eligibility:

People aged 15 to 17 years. Participants will come from urban, suburban, and rural areas in the United States. Factors such as race and gender will match US averages.

Participants will only include subjects recruited by Qualtrics from their national panel of available respondents, who have agreed to be contacted by Qualtrics with opportunities to participate in surveys.

Design:

Participants will be contacted by email. The email will include a link to the survey. The emails will be sent only to people who agreed to be contacted about taking surveys.

Participants will complete the survey online. It should take only 10 minutes.

Questions will include the following:

Have participants been vaccinated against COVID-19? Are they in the process of getting vaccinated?

Do they want to be vaccinated?

Have they had trouble getting vaccinated? If so, what kind of barriers did they face?

What reasons have they considered for and against getting vaccinated?

What have their personal experiences been with COVID-19?

What is their primary source of information about COVID-19?

Other questions will ask about:

Household size.

Employment of people in the household.

How many people in the house have been vaccinated.

The primary language spoken at home.

The natural history survey will be anonymous. Participants will not be asked to give their names....

DETAILED DESCRIPTION:
The project will survey a representative sample of US adolescents age 15-17 and English speaking. This age group has been selected because they are likely to currently be High School students and are eligible for vaccination under the current Emergency Use Authorization (EUA) for and approval of the Pfizer-BioNTech COVID vaccine. The Pfizer-BioNTech vaccine received an EUA for those 16 and over in December of 2020, and was approved for this age group in August of 2021. Pfizer received an EUA for those 12 to 15 in May of 2021.

We are targeting a total of 460 responses which will give us a sufficient sample size to have a target power of 0.901 and 0.05 alpha to test our primary hypothesis that adolescents in rural settings are more likely to have encountered barriers in their pursuit of COVID vaccination. The respondents will be a convenience sample recruited from the Qualtrics panel, with demographic characteristic quotas (race/ethnicity, gender etc..) to approximate the most recent US census. The inclusion criteria are: age 15-17, and living in urban, suburban or rural community

ELIGIBILITY:
* INCLUSION CRITERIA:
* age 15-17, and
* living in urban, suburban or rural community
* Participants will only include subjects recruited by Qualtrics from their national panel of available respondents, who have agreed to be contacted by Qualtrics with opportunities to participate in surveys.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We are collecting data from 15-17 year olds from US general population. Qualtrics will be retained to have access to sample.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Barriers Encountered | Once
  We will be asking 15-17 year olds if they encountered barriers when accessing COVID vaccination. Our primary outcome will be the number and types of barriers encountered.

SECONDARY OUTCOMES:
Reasons for and against vaccination | Once
  We will be asking 15-17 year olds about the reasons they considered for and against vaccination. Our primary outcome will be the number of reasons and ratio of for and against.

CONTACTS AND LOCATIONS:
Overall Officials: Holly A Taylor, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The survey will be anonymous.

REFERENCES:
- [Background] Middleman AB, Klein J, Quinn J. Vaccine Hesitancy in the Time of COVID-19: Attitudes and Intentions of Teens and Parents Regarding the COVID-19 Vaccine. Vaccines (Basel). 2021 Dec 21;10(1):4. doi: 10.3390/vaccines10010004. PMID 35062665
- [Background] Scherer AM, Gedlinske AM, Parker AM, Gidengil CA, Askelson NM, Petersen CA, Woodworth KR, Lindley MC. Acceptability of Adolescent COVID-19 Vaccination Among Adolescents and Parents of Adolescents - United States, April 15-23, 2021. MMWR Morb Mortal Wkly Rep. 2021 Jul 16;70(28):997-1003. doi: 10.15585/mmwr.mm7028e1. PMID 34264908